CLINICAL TRIAL: NCT00504309
Title: Omacor: Measures of Endothelial Function and triGlyceride Alteration
Brief Title: Vascular and Lipid Effects of Omega-3 Fatty Acids in People With Moderately Elevated Triglycerides
Acronym: OMEGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Reliant Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sheila G West, Professor of Biobehavioral Health, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: G214
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Hypertriglyceridemia
Keywords: triglycerides; hypertriglyceridemia; omega-3; n-3; eicosapentaenoic acid; EPA; docosahexaenoic acid; DHA; flow mediated dilation; fish; Moderate hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor; Fish Oils; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 4g P-OM3, then 1g P-OM3, then Placebo (Experimental): 4 g/day Dose Prescription Omega-3 acid ethyl esters (P-OM3)capsules(4) for first intervention (8 weeks), followed by 1g/day P-OM3 capsules(4) for 2nd intervention (8 weeks), followed by Placebo corn oil capsules, 4/day, for the 3rd intervention (8 weeks).
  Interventions: Drug: 4/day of 4g P-OM3 capsules; Drug: 4/day of 1g P-OM3 capsules; Drug: Corn Oil Placebo, 4 capsules/day for 8 weeks
- 1g P-OM3, then 4g P-OM3, then Placebo (Experimental): 1g capsules for 8-wks, followed by 6-wk washout. 4g capsules for 8 wks,followed by 6-wk washout. Placebo capsules for 8-wks.
  Interventions: Drug: 4/day of 4g P-OM3 capsules; Drug: 4/day of 1g P-OM3 capsules; Drug: Corn Oil Placebo, 4 capsules/day for 8 weeks
- Placebo, then 4g P-OM3, then 1g P-OM3 (Experimental): Corn Oil placebo capsules for 8-wks, followed by 6-wk washout. 4g P-OM3 capsules for 8-wks, followed by 6-wk washout. 1g P-OM3 for 8-wks.
  Interventions: Drug: 4/day of 4g P-OM3 capsules; Drug: 4/day of 1g P-OM3 capsules; Drug: Corn Oil Placebo, 4 capsules/day for 8 weeks
- 4g P-OM3, then Placebo, then 1g P-OM3 (Experimental): 4g capsules for 8-wks, followed by 6-wk washout. Placebo capsules for 8-wks, followed by 6-wk washout. 1g capsules for 8 wks.
  Interventions: Drug: 4/day of 4g P-OM3 capsules; Drug: 4/day of 1g P-OM3 capsules; Drug: Corn Oil Placebo, 4 capsules/day for 8 weeks
- 1g P-OM3, then Placebo, then 4g P-OM3 (Experimental): 1g capsules for 8-wks, followed by 6-wk washout. Placebo capsules for 8-wks, followed by 6-wk washout. 4g capsules for 8 wks.
  Interventions: Drug: 4/day of 4g P-OM3 capsules; Drug: 4/day of 1g P-OM3 capsules; Drug: Corn Oil Placebo, 4 capsules/day for 8 weeks
- Placebo, then 1g P-OM3, then 4g P-OM3 (Experimental): Corn oil placebo capsules for 8-wks, followed by 6-wk washout.1g capsules for 8-wks, followed by 6-wk washout. 4g capsules for 8 wks.
  Interventions: Drug: 4/day of 4g P-OM3 capsules; Drug: 4/day of 1g P-OM3 capsules; Drug: Corn Oil Placebo, 4 capsules/day for 8 weeks

INTERVENTIONS:
Drug: 4/day of 4g P-OM3 capsules — 4/day of 4g P-OM3 capsules for 8 weeks
  Other Names: OM3AEE; Lovaza; Fish oil
Drug: 4/day of 1g P-OM3 capsules — 4/day of 1g P-OM3 capsules for 8 weeks
  Other Names: OM3AEE; Lovaza; Fish oil
Drug: Corn Oil Placebo, 4 capsules/day for 8 weeks — 4 capsules per day of corn oil placebo for 8 weeks
  Other Names: Corn oil

SUMMARY:
The purpose of this study is to evaluate the cardiovascular and lipid effects of two doses of an omega-3 fatty acid concentrate in a group of people who normally are not treated for high lipids.

ELIGIBILITY:
Inclusion Criteria:

* triglycerides 150-500 mg/dL
* age 21-65 years
* generally healthy
* body mass index (BMI) 20-39 kg/m2

Exclusion Criteria:

* smoking
* premenopausal (if female)
* use of hormone replacement or oral contraceptives
* use of lipid lowering or blood pressure medication
* hypertension (blood pressure > 150/95 mm Hg)
* peripheral vascular disease
* heart disease, diabetes, or stroke
* inflammatory disease (e.g. rheumatoid arthritis or Crohn's)
* elevated liver enzymes
* high intake of omega-3 containing foods
* allergy to adhesive or latex
* use of aspirin, anticoagulants, or SSRI

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila G West, PhD, Principal Investigator — Penn State University; Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University; Ann C Skulas-Ray, B.S., Principal Investigator — Penn State University
Locations (1):
- Penn State University General Clinical Research Center, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Sauder KA, Skulas-Ray AC, Campbell TS, Johnson JA, Kris-Etherton PM, West SG. Effects of omega-3 fatty acid supplementation on heart rate variability at rest and during acute stress in adults with moderate hypertriglyceridemia. Psychosom Med. 2013 May;75(4):382-9. doi: 10.1097/PSY.0b013e318290a107. Epub 2013 Apr 16. PMID 23592752
- [Derived] Skulas-Ray AC, Kris-Etherton PM, Harris WS, West SG. Effects of marine-derived omega-3 fatty acids on systemic hemodynamics at rest and during stress: a dose-response study. Ann Behav Med. 2012 Dec;44(3):301-8. doi: 10.1007/s12160-012-9393-2. PMID 22865498
- [Derived] Skulas-Ray AC, Kris-Etherton PM, Harris WS, Vanden Heuvel JP, Wagner PR, West SG. Dose-response effects of omega-3 fatty acids on triglycerides, inflammation, and endothelial function in healthy persons with moderate hypertriglyceridemia. Am J Clin Nutr. 2011 Feb;93(2):243-52. doi: 10.3945/ajcn.110.003871. Epub 2010 Dec 15. PMID 21159789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4g P-OM3, Then 1g P-OM3, Then Placebo | 1g P-OM3, Then 4g P-OM3, Then Placebo | Placebo, Then 4g P-OM3, Then 1g P-OM3 | 4g P-OM3, Then Placebo, Then 1g P-OM3 | 1g P-OM3, Then Placebo, Then 4g P-OM3 | Placebo, Then 1g P-OM3, Then 4g P-OM3
Started | 7 | 5 | 2 | 3 | 8 | 3
Completed | 7 | 5 | 1 (Participant dropped out during second period) | 3 | 7 (Participant died during washout after 2nd period) | 3
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 subject in the "Placebo, 4 g P-OM3, 1 g P-OM3" sequence and 1 subject in the "1 g P-OM3, Placebo, 4 g P-OM3" sequence did not complete the study and were not included in the baseline analysis.
Groups:
- 4 g P-OM3, 1 g P-OM3, Placebo: 4 g/d prescription omega-3 fatty acid ethyl esters (P-OM3) for 8 weeks, followed by 1 g/d P-OM3 for 8 weeks, followed by 4 g/d corn oil placebo for 8 weeks
- 1 g P-OM3, 4 g P-OM3, Placebo: 1 g/d prescription omega-3 fatty acid ethyl esters (P-OM3) for 8 weeks, followed by 4 g/d P-OM3 for 8 weeks, followed by 4 g/d corn oil placebo for 8 weeks
- Placebo, 4 g P-OM3, 1 g P-OM3: 4 g/d corn oil placebo for 8 weeks, followed by 4 g/d prescription omega-3 fatty acid ethyl esters (P-OM3) for 8 weeks, followed by 1 g/d P-OM3 for 8 weeks
- 4 g P-OM3, Placebo, 1 g P-OM3: 4 g/d prescription omega-3 fatty acid ethyl esters (P-OM3) for 8 weeks, followed by 4 g/d corn oil placebo for 8 weeks, followed by 1 g/d P-OM3 for 8 weeks
- 1 g P-OM3, Placebo, 4 g P-OM3: 1 g/d prescription omega-3 fatty acid ethyl esters (P-OM3) for 8 weeks, followed by 4 g/d corn oil placebo for 8 weeks, followed by 4 g/d P-OM3 for 8 weeks
- Placebo, 1 g P-OM3, 4 g P-OM3: 4 g/d corn oil placebo for 8 weeks, followed by 1 g/d prescription omega-3 fatty acid ethyl esters (P-OM3) for 8 weeks, followed by 4 g/d P-OM3 for 8 weeks
- Total: Total of all reporting groups
Arm/Group | 4 g P-OM3, 1 g P-OM3, Placebo | 1 g P-OM3, 4 g P-OM3, Placebo | Placebo, 4 g P-OM3, 1 g P-OM3 | 4 g P-OM3, Placebo, 1 g P-OM3 | 1 g P-OM3, Placebo, 4 g P-OM3 | Placebo, 1 g P-OM3, 4 g P-OM3 | Total
Number analyzed (Participants) | 7 | 5 | 1 | 3 | 7 | 3 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 1 | 3 | 7 | 3 | 25
  >=65 years | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 2 | 0 | 3
  Male | 7 | 4 | 1 | 3 | 5 | 3 | 23
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 1 | 3 | 7 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Lipid Profile
Description: Plasma/serum samples were analyzed at baseline and at the end of each 8-week treatment period to evaluate the effect of P-OM3 dose on triglycerides, HDL-C, LDL-C, and total cholesterol.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- 4g P-OM3: 4 g/d Prescription Omega-3 acid ethyl esters (P-OM3)
- 1g P-OM3: 1 g/d Prescription Omega-3 acid ethyl esters (P-OM3)
- Placebo: 4 g/d corn oil placebo
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
mg/dL
  High density lipoprotein-cholesterol (HDL-C) | 43.2 (1.9) | 42.7 (1.9) | 42.6 (1.9)
  Low density lipoprotein-cholesterol (LDL-C) | 130.3 (7.6) | 127.6 (7.6) | 123.3 (7.6)
  Total Cholesterol | 207.9 (7.9) | 212.1 (7.9) | 209 (7.9)
  Triglycerides | 173.7 (17.5) | 215.3 (17.5) | 237.3 (17.5)
Statistical Analysis 1: Comparison: 4g P-OM3 vs 1g P-OM3 vs Placebo; Fasting triglycerides (mg/dL) were measured on two consecutive days and averaged for analysis at the end of each treatment period. The null hypothesis was that triglycerides did not differ between groups; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Tukey p-values were used for post hoc comparisons
Statistical Analysis 2: Comparison: 4g P-OM3 vs 1g P-OM3 vs Placebo; Cholesterol values were compared as the average of two fasting values at the end of each treatment. Cholesterol values included LDL-C, HDL-C, total cholesterol, and calculated ratios; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis

2. Primary Outcome: Flow-mediated Dilation (FMD)
Description: Effect of P-OM3 dose on FMD, which is measured as percent change in brachial artery diameter at peak dilation vs. baseline following a 5-minute occlusion period.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: % change in brachial artery diameter
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
% change in brachial artery diameter | 5.00 (0.5) | 4.03 (0.5) | 5.00 (0.5)

3. Primary Outcome: Blood Pressure
Description: Effect of P-OM3 dose on blood pressure
Time Frame: 8 weeks
Population: Two participants did not complete the study and were therefore excluded from analysis.
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- 4g P-OM3: 4 g Prescription Omega-3 acid ethyl esters (P-OM3)
- 1g P-OM3: 1 g Prescription Omega-3 acid ethyl esters (P-OM3)
- Placebo: Corn Oil Placebo
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
mm Hg
  Diastolic blood pressure (DBP) | 76.1 (1.6) | 77.7 (1.6) | 77.8 (1.6)
  Systolic blood pressure (SBP) | 126.3 (2.2) | 129.0 (2.2) | 128.4 (2.2)

4. Primary Outcome: Heart Rate
Description: Effect of P-OM3 dose on heart rate
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
beats per minute | 67.9 (1.8) | 69.8 (1.8) | 71.8 (1.8)

5. Secondary Outcome: Erythrocyte Fatty Acids
Description: Effect of P-OM3 dose on the percent concentration of select omega-3 fatty acids in red blood cells
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: percentage
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
percentage
  Eicosapentaenoic acid (EPA) | 2.30 (0.09) | 1.15 (0.09) | 0.57 (0.09)
  Docosahexaenoic acid (DHA) | 6.49 (0.15) | 5.34 (0.15) | 4.39 (0.15)
  Omega-3 Index (EPA + DHA) | 8.79 (0.21) | 6.49 (0.21) | 4.96 (0.21)

6. Secondary Outcome: Cytokine Inflammatory Markers
Description: Effect of P-OM3 dose on concentrations of circulating inflammatory markers in plasma
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
pg/mL
  Interleuken-1β (IL-1β) | 0.14 (0.02) | 0.15 (0.02) | 0.15 (0.02)
  Interleuken-6 (IL-6) | 0.87 (0.15) | 0.85 (0.15) | 0.87 (0.15)
  Tumor Necrosis Factor-α (TNF-α) | 1.00 (0.07) | 1.11 (0.14) | 1.20 (0.14)

7. Secondary Outcome: Fasting Glucose
Description: Effect of P-OM3 dose on fasting glucose
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
mg/dL | 99.2 (1.9) | 98.0 (1.9) | 96.1 (2.0)

8. Secondary Outcome: Psychosocial Profile Questionnaires
Description: Effect of P-OM3 dose on psychosocial questionnaires:
  Perceived Stress Scale (PSS)
  * 14 questions, scored 0-4 based on how often the subject felt certain emotions
  * Scores: 0 to 40; higher scores indicate higher perceived stress
  Spielberger State Anxiety Inventory
  * Levels of state anxiety (situational) and trait anxiety; 40 items scored by a Likert scale
  * Scores: 20 to 80; higher scores indicate higher levels of anxiety
  Positive and Negative Affect Scales (PANAS)
  * Two 10-item scales; each item is rated on a Likert scale of 1 (not at all) to 5 (very much).
  * Scores: 10 to 50, with higher scores representing higher levels of positive or negative affect
  Center for Epidemiologic Studies Depression (CES-D) Scale
  * 20 questions about symptoms of depression in the past week
  * Scores: 0 to 60; higher scores indicate more symptomology. Score of 16 or higher indicates a risk for depression and should be followed by further evaluation by a qualified health professional
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
scores on a scale
  Perceived Stress Scale (PSS) | 23.2 (2.2) | 23.7 (2.4) | 22.3 (2.3)
  Positive Scale (PANAS) | 34.1 (2.2) | 35.0 (2.4) | 35.2 (2.3)
  Negative Scale (PANAS) | 11.7 (2.4) | 13.3 (2.5) | 11.9 (2.4)
  CES-D | 3.4 (2.9) | 3.3 (3.1) | 2.2 (3.0)
  Spielberger State Anxiety Inventory | 46.2 (1.5) | 46.5 (1.6) | 45.0 (1.6)

9. Secondary Outcome: C-reactive Protein (CRP)
Description: Effect of P-OM3 dose on the plasma concentration of the inflammatory marker CRP
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
mg/L | 1.29 (0.2) | 1.32 (0.2) | 1.45 (0.2)

10. Secondary Outcome: Fasting Insulin
Description: Effect of P-OM3 dose on fasting insulin
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: μIU/mL
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
μIU/mL | 15.0 (1.4) | 15.5 (1.4) | 14.6 (1.4)

11. Secondary Outcome: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) and Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: Effect of P-OM3 dose on the homeostatic model assessment of insulin resistance (HOMA-IR) and the quantitative insulin sensitivity check index (QUICKI).
  HOMA-IR calculates an index of insulin resistance and is calculated as follows: HOMA-IR = (glucose mg/dL * insulin mU/L) / 405.
  QUICKI is calculated as follows: QUICKI = 1 / (log(fasting insulin µU/mL) + log(fasting glucose mg/dL)).
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: index units
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Number analyzed (Participants) | 26 | 26 | 26
index units
  HOMA-IR | 3.64 (0.4) | 3.75 (0.4) | 3.55 (0.4)
  QUICKI | 0.14 (0.002) | 0.14 (0.002) | 0.14 (0.002)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected while participants were enrolled (approximately 2.5 years).
Arm/Group | 4g P-OM3 | 1g P-OM3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 1/27 | 0/27 | 0/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4g P-OM3 (N=27) | 1g P-OM3 (N=27) | Placebo (N=28)
Gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Lower GI symptoms that contributed to withdrawal from the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No